CLINICAL TRIAL: NCT01256489
Title: Infliximab Therapy to Improve Retention of the Boston Keratoprosthesis in Patients After Stevens Johnson Syndrome/ Toxic Epidermal Necrolysis
Brief Title: Infliximab to Improve Retention of the Boston Keratoprosthesis in Patients After Stevens Johnson Syndrome/ Toxic Epidermal Necrolysis (SJS/TENS)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Steven Johnson's Syndrome (SJS) and Toxic Epidermal Necrolysis Syndrome (TENS) are rare (~3 in 1 million). No eligible subjects have been identified.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-02-010; 196405 (Other: MEEI Human Studies Committee)
Record Dates: First submitted 2010-11-19; First posted 2010-12-08 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-01

CONDITIONS: Stevens-Johnson Syndrome; Corneal Blindness
Keywords: KPro; Keratoprosthesis; Stevens-Johnson Syndrome; Infliximab; Corneal Blindness
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infliximab (Other): Every patient enrolled in the study will receive monthly infusions of Infliximab throughout the term of the study. Infliximab will be administered intravenously.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — The drug will be administered intravenously every month for 110 weeks (duration of the study). The initial dose of infliximab will be 5mg/kg of body weight. The dose may be adjusted up to a maximal dosing of 10mg/kg depending upon disease activity, as judged by the investigators.
  Other Names: Remicade

SUMMARY:
The proposed study is intended to test the idea, based upon current knowledge of the biology and physiology of corneal ulceration in SJS/TENS patients who receive a keratoprosthesis, and on the known effects of infliximab on matrix metalloproteinases, that infliximab therapy for such patients may reduce the likelihood of corneal ulceration, and hence extend the period of prosthesis retention and vision recovery.

DETAILED DESCRIPTION:
The closely related disorders, Stevens Johnson Syndrome (SJS) and Toxic Epidermal Necrolysis Syndrome (TENS), represent rare but severe hypersensitivity responses to a systemic medication, and cause severe sloughing of the skin and mucous membranes. Approximately half of affected patients experience ocular involvement, which can lead to corneal opacity and vascularization, and in some patients, blindness. Corneal transplantation (corneal allograft) is typically unsuccessful in SJS/TENS, because of chronic inflammation at the ocular surface, leading to corneal neovascularization and opacity, tissue melt, ulceration, and perforation.

The Boston keratoprosthesis, an artificial cornea developed at the Massachusetts Eye and Ear Infirmary (MEEI) over the last 40 years, is an FDA approved device for patients with corneal blindness not amenable to corneal transplantation, and has restored the sight of thousands of such patients, but in SJS/TENS patients remains associated with tissue melts (tissue ulceration), perforation, and ultimately in some, loss of the eye. K-Pro surgery is currently the best option for patients with SJS or TENS and corneal blindness, but these patients also have the worst prognosis after surgery. While the outcomes of these surgeries for patients with SJS or TENS have improved dramatically in the past ten years, they are still unsatisfactory. Remicade® has been used in a small group of patients with SJS or TENS undergoing K-Pro surgery, with one remarkable success. The purpose of this study is to explore this treatment more fully.

For a case report detailing the use of infliximab in one patient, see the following article: Dohlman JG, Foster CS, Dohlman CH. "Boston Keratoprosthesis in Stevens-Johnson Syndrome: A case of using infliximab to prevent tissue necrosis." Digital Journal of Ophthalmology. 2009, Volume 15, Number 1.

Recently developed biologics have dramatically improved functional outcomes and quality of life in patients with autoimmune diseases. One such agent, infliximab, acts by blocking TNF alpha, a protein associated with tissue melting in the cornea, and is increasingly being used for autoimmune eye conditions, in addition to its FDA approved indication for recalcitrant rheumatoid arthritis.

The proposed study will determine the feasibility of combining infliximab with keratoprosthesis surgery, and will closely monitor patients for episodes of corneal melting: the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy proven SJS/TENS with corneal opacity and neovascularization
* Bilateral legal blindness (<20/200 in better eye)
* 18 years of age or older
* Able to provide informed consent
* Sufficiently healthy to undergo infliximab infusions, surgery, and a vigorous postoperative follow-up course
* Able to administer eye medications or have a care giver able and willing to do same
* Are considered eligible according to the following tuberculosis (TB) screening criteria:

  * Have no history of latent or active TB prior to screening.
  * Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
  * Have had no recent close contact with a person with active TB.
  * Within 6 weeks prior to the first administration of study agent, have a negative QuantiFERON-TB Gold test result (see Attachment A). Indeterminate results should be handled as outlined in the Screening Visit Section. A negative tuberculin skin test is considered acceptable if the QuantiFERON- TB Gold test is not acceptable in that country.
  * Have a chest radiograph (posterior-anterior view) taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current, active TB or old, inactive TB.

Exclusion Criteria:

* Visual acuity >20/200 in better eye
* Corneal blindness not due to effects of SJS/TENS
* Hypersensitivity to infliximab or chemically related medication
* Pregnant or lactating
* Have a history of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, prior to screening. Refer to inclusion criteria for information regarding eligibility with a history of latent TB.
* Have had a Bacille Calmette-Guérin (BCG) vaccination within 12 months of screening.
* Have a chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of a malignancy or current active infection, including TB.
* Have had a nontuberculous mycobacterial infection or opportunistic infection (eg, cytomegalovirus, pneumocystosis, aspergillosis) within 6 months prior to screening.
* Have indeterminate initial and repeat QuantiFERON-TB Gold test results.
* History or current diagnosis of diabetes mellitus
* History of immune system problem other than Stevens Johnson Syndrome
* History of recurrent infections
* History or current diagnosis of cancer
* Active psoriasis
* History of heart failure
* History of hepatitis B virus
* MRSA or VRE infection
* Nervous system disorders such as multiple sclerosis or Guillain-Barre syndrome
* Scheduled to receive a live vaccine at any time point during study participation
* Currently receiving treatments of Kineret (Anakinra)
* Unable to attend postoperative visits or administer medications, or no care giver available and willing to assist with same

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of corneal ulceration | Assessed monthly for up to 2 years following surgery

SECONDARY OUTCOMES:
Occurrence of systemic adverse events | Assessed monthly for up to 2 years following first infusion
Period Of Prosthesis Retention | Assessed monthly for up to 2 years following surgery
Vision Recovery | Assessed monthly for up to 2 years following surgery

CONTACTS AND LOCATIONS:
Overall Officials: James Chodosh, MD, MPH, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States